CLINICAL TRIAL: NCT07317128
Title: Study to Evaluate the Efficacy of Two Occlusion Technology Dentifrices in the Relief of Dentinal Hypersensitivity
Brief Title: Study to Evaluate the Effectiveness of Test Dentifrice in the Relief of Dentinal Hypersensitivity
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: HALEON (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: RH01748
Record Dates: First submitted 2025-12-19; First posted 2026-01-05 (Actual); Last update posted 2026-01-05 (Actual); Status verified 2025-12

CONDITIONS: Dentin Sensitivity
MeSH Terms: conditions — Dentin Sensitivity

STUDY DESIGN:
Who Masked: Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Test Dentifrice (Experimental): Participants will be instructed to apply a full ribbon of test dentifrice to cover the head of the assigned toothbrush and brush twice daily for 1 timed minute throughout the 12-week treatment period.
  Interventions: Drug: Test Dentifrice
- Comparator Dentifrice (Active Comparator): Participants will be instructed to apply a full ribbon of the comparator dentifrice to cover the head of the assigned toothbrush and brush twice daily for 1 timed minute throughout the 12-week treatment period.
  Interventions: Drug: Colgate Sensitive ProRelief
- Negative Control Dentifrice (Active Comparator): Participants will be instructed to apply a full ribbon of the negative control dentifrice to cover the head of the assigned toothbrush and brush twice daily for 1 timed minute throughout the 12-week treatment period.
  Interventions: Drug: Colgate Triple Protection

INTERVENTIONS:
Drug: Test Dentifrice — Dentifrice containing 1450 parts per million (ppm) fluoride as sodium monofluorophosphate.
  Arms: Test Dentifrice
Drug: Colgate Sensitive ProRelief — A marketed dentifrice.
  Arms: Comparator Dentifrice
Drug: Colgate Triple Protection — A marketed dentifrice.
  Arms: Negative Control Dentifrice

SUMMARY:
The purpose of this study is to compare the clinical efficacy of test fluoride dentifrice in reducing Dentin Hypersensitivity (DH) with that of a standard fluoride dentifrice, as measured by evaporative air sensitivity after 12 weeks twice daily brushing.

DETAILED DESCRIPTION:
A randomized, examiner blind, three treatment arm, parallel group design with a treatment period of 12 weeks. Approximately 275 participants will be screened to ensure that approximately 120 participants to be randomized (approximately 40 to each treatment group) and at least 114 participants to complete the study (approximately 38 per treatment group).

ELIGIBILITY:
Inclusion Criteria:

* Participant demonstrates understanding of the study and is willing to participate as evidenced by voluntary written informed consent and has received a signed and dated copy of the informed consent form.
* Participant is 18 to 60 years of age.
* Participant understands and is willing, able and likely to comply all study procedures and restrictions.
* Participant with good general and mental health, in the opinion of the investigator or medically qualified designee:

  1. No clinically significant and relevant abnormalities of medical history or physical /oral examination.
  2. Absence of any condition that would impact on the participant's safety or wellbeing or affect the participant's ability to understand and follow study procedures and requirements.
* Self-reported history of DH lasting more than 6 months but not more than 10 years and minimum of 20 natural teeth.

Exclusion Criteria:

* Female participant who is known to be pregnant or who is intending to become pregnant over the duration of the study.
* Female participant who is breast-feeding.
* Participant with known or suspected intolerance or hypersensitivity to the study materials (or closely related compounds) or any of their stated ingredients.
* Participation is in another clinical study or receipt of an investigational drug within 30 days prior to the screening visit.
* Participant who has had tooth desensitizing treatment within 8 weeks of Screening visit (professional sensitivity treatments and non-dentifrice sensitivity treatments).
* Participant who had previously participated in this study.
* Participant with a recent history (within the last year) of alcohol or other substance abuse.
* Participant who is an employee of the sponsor or the study site or members of their immediate family.
* Participant with presence of chronic debilitating disease which, in the opinion of the investigator, could affect study outcomes.
* Participant with any condition or daily doses of a medication which, in the opinion of the investigator, is causing xerostomia.
* Participant with dental prophylaxis within 4 weeks of screening.
* Participant with tongue or lip piercing or presence of dental implants.
* Participant with gross periodontal disease, treatment of periodontal disease (including surgery) within 12 months of screening, scaling or root planning within 3 months of screening.
* Participant who did teeth bleaching within 8 weeks of screening.
* Participant with Specific Dentition Exclusions for Test teeth.

  1. Tooth with evidence of current or recent caries, or reported treatment of decay in 12 months of screening.
  2. Tooth with exposed dentine but with deep, defective or facial restorations, teeth used as abutments for fixed or removable partial dentures, teeth with full crowns or veneers, orthodontic bands or cracked enamel. Sensitive teeth with contributing aetiologies other than erosion, abrasion or recession of exposed dentine.
  3. Sensitive teeth are not expected, in the opinion of the investigator, to respond to treatment with an over-the-counter dentifrice.
* Participant who has used product of a sensitivity dentifrice within 8 weeks of screening.
* Participant who had daily doses of a medication or traditional herbal ingredients or treatments which, in the opinion of the investigator, could interfere with the perception of pain. Examples of such medications include analgesics, anticonvulsants, antihistamines that cause marked or moderate sedation, sedatives, tranquilizers, mood-altering and anti-inflammatory drugs. Examples of herbal ingredients/treatments include clove oil, olive oil, or other treatments that are directly applied to the oral cavity for the treatment of oral health problems.
* Participant who is currently taking a course of antibiotics or has taken a course of antibiotics within 2 weeks of baseline.
* Participant who had dental procedures or participant who require antibiotic prophylaxis for dental procedures.
* Any participant who, in the opinion of the investigator, should not participate in the study.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 120 (Actual)
Dates: Start 2013-01-20 (Actual); Primary Completion 2013-06-08 (Actual); Study Completion 2013-06-08 (Actual)

PRIMARY OUTCOMES:
Change from Baseline in Schiff Sensitivity Score at Week 12 (Test Dentifrice Versus [vs] Negative Control Dentifrice) | Baseline and Week 12
  Evaporative (air) sensitivity is evaluated using the Schiff Sensitivity Score on test teeth for each participant. After the examiner applies a standardized air stimulus, the participant's response is rated on a 0 to 3 scale, where 0= no response to the stimulus, 1= response to air stimulus without request for discontinuation of the stimulus, 2= response to air stimulus with request for discontinuation of the stimulus, and 3= a painful response with a request for discontinuation of the stimulus. The lower score indicates improvement. Change from baseline will be calculated by subtracting the baseline score from the score at Week 12.

SECONDARY OUTCOMES:
Change from Baseline in Schiff Sensitivity Score at Weeks 2, 4 and 8 (Test Dentifrice vs Negative Control Dentifrice) | Baseline, Weeks 2, 4, and 8
  Evaporative (air) sensitivity is evaluated using the Schiff Sensitivity Score on test teeth for each participant. After the examiner applies a standardized air stimulus, the participant's response is rated on a 0 to 3 scale, where 0= no response to the stimulus, 1= response to air stimulus without request for discontinuation of the stimulus, 2= response to air stimulus with request for discontinuation of the stimulus, and 3= a painful response with a request for discontinuation of the stimulus. The lower score indicates improvement. Change from baseline will be calculated by subtracting the baseline score from the score at the indicated timepoints.
Mean Change from Baseline in Visual Analogue Scale (VAS) at Weeks 2, 4, 8 and 12 (Test Dentifrice vs Negative Control Dentifrice) | Baseline, Weeks 2, 4, 8 and 12
  Evaporative (air) sensitivity is assessed on the test teeth by applying a 1-second air stimulus from a standard dental syringe. Participants will rate the intensity of their response to the evaporative (air) stimulus using a 100 millimeter (mm) VAS with scores ranging from 0 mm (No discomfort) to 100 mm (Extreme discomfort; worst imaginable). Higher score indicates worse outcome (higher sensitivity). Change from Baseline will be calculated by subtracting Baseline value from the value at indicated timepoints.
Mean Change from Baseline in Tactile Threshold at Weeks 2, 4, 8 and 12 (Test Dentifrice vs Negative Control Dentifrice) | Baseline, Weeks 2, 4, 8 and 12
  Tactile sensitivity is assessed for eligible teeth using a constant pressure probe (Yeaple probe). After each application of the stimulus, the participant will be asked to indicate whether they experienced any pain or discomfort (yes/no response). The pressure setting with two consecutive 'yes' responses will be recorded as the tactile threshold (grams [g]). Higher tactile threshold indicates better outcome (less sensitivity). Change from Baseline will be calculated by subtracting Baseline value from the value at indicated timepoints.
Mean Change from Baseline in Schiff Sensitivity Score at Weeks 2, 4, 8 and 12 (Comparator Dentifrice vs Negative Control Dentifrice) | Baseline, Weeks 2, 4, 8 and 12
  Evaporative (air) sensitivity is evaluated using the Schiff Sensitivity Score on test teeth for each participant. After the examiner applies a standardized air stimulus, the participant's response is rated on a 0 to 3 scale, where 0= no response to the stimulus, 1= response to air stimulus without request for discontinuation of the stimulus, 2= response to air stimulus with request for discontinuation of the stimulus, and 3= a painful response with a request for discontinuation of the stimulus. The lower score indicates improvement. Change from baseline will be calculated by subtracting the baseline score from the score at the indicated timepoints.
Mean Change from Baseline in VAS at Weeks 2, 4, 8 and 12 (Comparator Dentifrice vs Negative Control Dentifrice) | Baseline, Weeks 2, 4, 8 and 12
  Evaporative (air) sensitivity is assessed on the test teeth by applying a 1-second air stimulus from a standard dental syringe. Participants will rate the intensity of their response to the evaporative (air) stimulus using a 100 mm VAS with scores ranging from 0 mm (No discomfort) to 100 mm (Extreme discomfort; worst imaginable). Higher score indicates worse outcome (higher sensitivity). Change from Baseline will be calculated by subtracting Baseline value from the value at indicated timepoints.
Mean Change from Baseline in Tactile Threshold at Weeks 2, 4, 8 and 12 (Comparator Dentifrice vs Negative Control Dentifrice) | Baseline, Weeks 2, 4, 8 and 12
  Tactile sensitivity is assessed for eligible teeth using a constant pressure probe (Yeaple probe). After each application of the stimulus, the participant will be asked to indicate whether they experienced any pain or discomfort (yes/no response). The pressure setting with two consecutive 'yes' responses will be recorded as the tactile threshold (g). Higher tactile threshold indicates better outcome (less sensitivity). Change from Baseline will be calculated by subtracting Baseline value from the value at indicated timepoints.
Mean Change from Baseline in Schiff Sensitivity Score at Weeks 2, 4, 8 and 12 (Test Dentifrice vs Comparator Dentifrice) | Baseline, Weeks 2, 4, 8 and 12
  Evaporative (air) sensitivity is evaluated using the Schiff Sensitivity Score on test teeth for each participant. After the examiner applies a standardized air stimulus, the participant's response is rated on a 0 to 3 scale, where 0= no response to the stimulus, 1= response to air stimulus without request for discontinuation of the stimulus, 2= response to air stimulus with request for discontinuation of the stimulus, and 3= a painful response with a request for discontinuation of the stimulus. The lower score indicates improvement. Change from baseline will be calculated by subtracting the baseline score from the score at the indicated timepoints.
Mean Change from Baseline in VAS at Weeks 2, 4, 8 and 12 (Test Dentifrice vs Comparator Dentifrice) | Baseline, Weeks 2, 4, 8 and 12
  Evaporative (air) sensitivity is assessed on the test teeth by applying a 1-second air stimulus from a standard dental syringe. Participants will rate the intensity of their response to the evaporative (air) stimulus using a 100 mm VAS with scores ranging from 0 mm (No discomfort) to 100 mm (Extreme discomfort; worst imaginable). Higher score indicates worse outcome (higher sensitivity). Change from Baseline will be calculated by subtracting Baseline value from the value at indicated timepoints.
Mean Change from Baseline in Tactile Threshold at Weeks 2, 4, 8 and 12 (Test Dentifrice vs Comparator Dentifrice) | Baseline, Weeks 2, 4, 8 and 12
  Tactile sensitivity is assessed for eligible teeth using a constant pressure probe (Yeaple probe). After each application of the stimulus, the participant will be asked to indicate whether they experienced any pain or discomfort (yes/no response). The pressure setting with two consecutive 'yes' responses will be recorded as the tactile threshold (g). Higher tactile threshold indicates better outcome (less sensitivity). Change from Baseline will be calculated by subtracting Baseline value from the value at indicated timepoints.

CONTACTS AND LOCATIONS:
Overall Officials: Minquan Du, DSS, PhD, Principal Investigator — Wuhan University
Locations (1):
- School and Hospital of Stomatology, Wuhan University, Wuhan, Hubei, China

IPD SHARING:
Plan to Share IPD: Yes
Anonymized individual participant data and study documents can be requested for further research from ww.clinical-trial-register@haleon.com.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: IPD will be made available within 6 months of publishing the results of the primary endpoints, key secondary endpoints and safety data of the study.
Access Criteria: Access is provided after a research proposal is submitted and has received approval from the Independent Review Panel and after a Data Sharing Agreement is in place. Access is provided for an initial period of 12 months, but an extension can be granted, when justified, for up to another 12 months.